CLINICAL TRIAL: NCT06809621
Title: A Study Investigating the Pharmacokinetic and Pharmacodynamic Properties and Safety and Tolerability of NNC0471-0119 H When Administered as Bolus in a Continuous Subcutaneous Insulin Infusion Regimen in Participants With Type 1 Diabetes
Brief Title: A Study to Test How Insulin NNC0471-0119 H Works in the Body in Participants With Type 1 Diabetes When Given by an Insulin Pump
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1471-7712; U1111-1306-8005 (Other: World Health Organization (WHO)); 2024-513472-18 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC0471-0119 H then Insulin Aspart (Experimental): Participants will receive NNC0471-0119 H subcutaneously (s.c.) in period 1 followed by insulin aspart s.c. in period 2.
  Interventions: Drug: NNC0471-0119 H; Drug: Insulin aspart
- Insulin Aspart then NNC0471-0119 H (Active Comparator): Participants will receive insulin aspart s.c. in period 1 followed by s.c. NNC0471-0119 H in period 2.
  Interventions: Drug: NNC0471-0119 H; Drug: Insulin aspart

INTERVENTIONS:
Drug: NNC0471-0119 H — NNC0471-0119 H will be administered subcutaneously.
Drug: Insulin aspart — Insulin aspart will be administered subcutaneously.

SUMMARY:
The study is looking at the effect and safety of a new fast-acting insulin (NNC0471 0119) to people with type 1 diabetes when given by an insulin pump. The study tests how fast insulin NNC0471-0119 enters your bloodstream, how long it stays there and how much it lowers blood sugar. The new insulin NNC0471-0119 will be compared to insulin aspart. The participants will get each study medicine administered at separate clinic visits. The study will last for about 1-3 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-64 years (both inclusive) at the time of signing the informed consent.
* Diagnosed with Type 1 Diabetes (T1D) greater than or equal to (≥) 1 year before screening.
* Insulin administration using continuous subcutaneous insulin infusion via a pump greater than or equal to (≥) 90 days before screening.
* Current daily insulin treatment between 0.2 and 1.2 Insulin units per kilogram per day [(I)U/kg/day] (both inclusive).

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
AUC(GIR,0-1h,basal-corrected): Area under the basal-corrected glucose infusion rate (GIR)-time curve from 0 to 1 hour | 0 to 1 hour after bolus infusion
  Measured in milligram per kilogram (mg/kg).

SECONDARY OUTCOMES:
AUC(GIR,0-t,basal-corrected): Area under the basal-corrected GIR-time curve from 0 to t | 0 to 9 hours after bolus infusion
  Measured in milligram per kilogram (mg/kg).
AUC(GIR,0-1h,basal-corrected)/AUC(GIR,0-t,basalcorrected):Ratio of the area under the basal-corrected GIR-time curve from 0 to 1 hour and 0 to t | 0 to 9 hours after bolus infusion
  Measured in percentage (%).
GIR(max,basal-corrected): Maximum observed basal-corrected GIR | 0 to 9 hours after bolus infusion
  Measured in milligrams per kilogram *minute (mg/[kg*min]).
AUC(NNC0471-0119,0-30min,basal corrected)/AUC(NNC0471-0119,0-t,basal-corrected):Ratio of basal-corrected area under serum NNC0471-0119 conc. time curve from 0-30min and 0-t | 0 to 9 hours after bolus infusion
  Measured in percentage (%).
AUC(NNC0471-0119,0-t,basal-corrected): Area under the basal-corrected serum NNC0471-0119 concentration time curve from 0 to t | 0 to 9 hours after bolus infusion
  Measured in hours*picomole per liter (h*pmol/L).
AUC(NNC0471-0119,0-30min,basal-corrected): Area under the basal-corrected serum NNC0471-0119 concentration time curve from 0 to 30 minutes | 0 to 30 minutes after bolus infusion
  Measured in h*pmol/L.
AUC(NNC0471-0119,2h-t,basal-corrected): Area under the basal-corrected serum NNC0471-0119 concentration time curve from 2 hours to t, where t is the first time the curve is back to basal level after bolus infusion (at most 9 hours) | 2 to 9 hours after bolus infusion
  Measured in h*pmol/L.
AUC(NNC0471-0119,2h-t,basal-corrected)/AUC(NNC0471-0119 H,0-t,basal-corrected):Ratio of basal corrected area under serum NNC0471-0119 conc. time curve from 2hrs-t and 0-t | 0 to 9 hours after bolus infusion
  Measured in percentage (%).
C(max,NNC0471-0119,basal-corrected): Maximum observed basal-corrected serum NNC0471-0119 concentration | 0 to 9 hours after bolus infusion
  Measured in picomoles per litre (pmol/L).
t(early50%Cmax,NNC0471-0119,basal-corrected): Time to early 50% maximum observed basal-corrected serum NNC0471-0119 concentration | 0 to 9 hours after bolus infusion
  Measured in minutes (Min).
t(late50%Cmax,NNC0471-0119,basal-corrected): Time to late 50% maximum observed basal-corrected serum NNC0471-0119 concentration | 0 to 9 hours after bolus infusion
  Measured in minutes (Min).
Number of adverse events (AEs) | From start of first investigational medicinal product (IMP) basal rate infusion (Visit 2, day -1) until completion of post-treatment end of study visit (Visit 4)
  Measure in number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com